CLINICAL TRIAL: NCT03080922
Title: Treatment of Relapsed/Refractory Acute Myeloblastic Leukemia(AML) by Infusion of Donor High Dose Allogeneic Mismatched Hematopoietic Stem Cells After Chemotherapy
Brief Title: High Dose Donor Hematopoietic Stem Cell Infusion for Relapsed/Refractory AML
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: The Affiliated Hospital of the Chinese Academy of Military Medical Sciences (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HD-DSI-AML
Record Dates: First submitted 2017-03-10; First posted 2017-03-15 (Actual); Last update posted 2017-04-04 (Actual); Status verified 2017-03

CONDITIONS: Leukemia, Myeloid
Keywords: Acute Myeloid Leukemia; Relapsed; Refractory; hematopoietic stem cell
MeSH Terms: conditions — Leukemia, Myeloid; Leukemia, Myeloid, Acute; Recurrence

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- hematopoietic stem cell (Experimental): high dose of donor granulocyte colony-stimulating factor（G-CSF）mobilized peripheral blood hematopoietic stem cell are infused to patient received normal chemotherapy
  Interventions: Biological: hematopoietic stem cell

INTERVENTIONS:
Biological: hematopoietic stem cell — high dose of donor G-CSF mobilized peripheral blood hematopoietic stem cell are infused to patient received normal chemotherapy

SUMMARY:
The purpose of this study is to evaluate the safety and efficiency of high dose allogeneic mismatched hematopoietic stem cells infusions after normal chemotherapy in patients with relapsed/refractory acute myeloid leukemia（AML）.

DETAILED DESCRIPTION:
The relapsed/refractory AML patients will receive IA/DA/MA(I,Idamycin，D，Daunorubicin，M，Mitoxantrone，A，cytosine arabinoside) chemotherapy followed by infusion of high dose allogeneic mismatched hematopoietic stem cells.

no graft-versus-host disease (GVHD) prevention will be conducted before transplantation. Cytokine storm,GVHD snd donor graft will be detected post-transplantation.

ELIGIBILITY:
Inclusion Criteria:

* Patient with relapsed and/or refractory AML
* Estimated life expectancy ≥ 12 weeks (according to investigator's judgment)
* Eastern Cooperative Oncology Group (ECOG) performance status ≤ 2

Exclusion Criteria:

* Previous treatment with investigational gene or cell therapy medicine products
* Any uncontrolled active medical disorder that would preclude participation as outlined

Ages: 15 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2016-03 (Actual); Primary Completion 2018-03 (Estimated); Study Completion 2019-03 (Estimated)

PRIMARY OUTCOMES:
complete remission rate | 2 months

SECONDARY OUTCOMES:
Disease-free survival | 2 years
Overall survival | 2 years
donor graft rate | 6 months
Occurrence of study related adverse events | 6 months
  defined as >= Grade 3 signs/symptoms, laboratory toxicities, and clinical events) that are possibly, likely, or definitely related to study treatment

CONTACTS AND LOCATIONS:
Overall Officials: HUISHENG AI, Study Chair — Affiliated Hospital of Academy of Military Medical Sciences
Locations (1):
- Affiliated Hospital of Academy of Military Medical Sciences ,, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided